CLINICAL TRIAL: NCT04479111
Title: An Open, Single-arm, Single Center, Clinical Trial to Investigate the Feasibility and Safety of Laparoscopic Ileocecus-sparing Right Hemicolectomy for Cancer of the Hepatic Flexure and Proximal Transverse Colon
Brief Title: Laparoscopic IIeocecus-Sparing Right Hemicolectomy for Cancer of the Hepatic Flexure and Proximal Transverse Colon
Acronym: LISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCCZ-S02
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hepatic Flexure Colon Cancer; Proximal Transverse Colon Cancer
Keywords: hepatic flexure colon cancer; proximal transverse colon cancer; ileocecus-sparing; laparoscopic right hemicolectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LISRH group (Experimental): Following the principle of complete mesocolic excision(CME), Ileocecus-Sparing Right colectomy refers to the resection of the most portion of the ascending colon, hepatic flexure and mid to distal transverse colon. The extent of lymph node dissection and length of distal resection margin are similar to conventional right hemicolectomy. The length of proximal resection margin varies.
  Interventions: Procedure: laparoscopic ileocecus-sparing right hemicolectomy

INTERVENTIONS:
Procedure: laparoscopic ileocecus-sparing right hemicolectomy — The ileocecal artery(ICA) is skeletonized. The colic branch of ICA is divided and ligated. Preserve anterior cecal artery, posterior cecal artery and ileocecal branch of ICA. Divide and ligate the right colic artery(RCA) and middle colic artery(MCA) at their roots. Dissect the lymph nodes surrounding the ICA, RCA and MCA accordingly. Head-to-Head colocolic anastomois is done, with circular stapler via making an opening at the bottom of cecum.

SUMMARY:
To investigate whether laparoscopic ileocecus-sparing right hemicolectomy is feasible and oncologically safe

DETAILED DESCRIPTION:
Our study is a single arm, single center clinical trial. The enrolled patients will accept laparoscopic ileocecus-sparing right hemicolectomy. The primary endpoint: postoperative complications, 1-year local recurrence. The second endpoint: conversion to conventional right hemicolectomy, time to first flatus after surgery, number of harvested lymph nodes, 3-year disease free survival, R0 resection, Specimen morphometry

ELIGIBILITY:
Inclusion Criteria:

1. Patients suitable for curative surgery 18-75years old
2. ASA grade I-III
3. Qualitative diagnosis: a pathological diagnosis of adenocarcinoma;
4. Localization diagnosis: the tumor located at hepatic flexure and proximal transverse colon(proximal to the right branch of middle colic artery);
5. Enhanced CT scan of chest, abdominal and pelvic cavity: assessment of tumor stage is T1-T4N0 or TanyN+; there is no distant metastasis.
6. Intraoperative measurement: the distance between colic branch of ileocolic artery and proximal edge of the tumor should be longer than 5cm.
7. Informed consent

Exclusion Criteria:

1. Simultaneous or metachronous multiple primary colorectal cancer;
2. History of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.
3. Preoperative imaging examination results show: fused lymph node at the root of ileocolic artery.
4. Distant metastasis.
5. History of any other malignant tumor in recent 5 years.
6. Patients need emergency operation.
7. Not suitable for laparoscopic surgery (i.e., extensive adhesion caused by abdominal surgery, not suitable for artificial pneumoperitoneum, etc).
8. Informed consent refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | up to 90 days after surgery
  Postoperative complications used to calculate the Comprehensive Complication Index (CCI) will be recorded
1-year local recurrence | 7 days after surgery
  rate of local recurrence one year after surgery, including anastomotic recurrence, recurrence around ileocolic vessels and surgical trunk of superior mesenteric vein,

SECONDARY OUTCOMES:
Conversion to conventional right hemicolectomy | 1 day of surgery
  the rate of conversion to conventional right hemicolectomy
Time to first flatus after surgery | up to 7 days after surgery
  days from a colectomy procedure to first occurrence of flatus during subject's postoperative recovery
Number of harvested lymph nodes | up to 1 week after surgery
  Number of harvested Lymph nodes according to the pathological report
R0 resection | up to 1 week after surgery
  Rate of resection without any affected margins during the surgical procedure according to the pathological report
Specimen morphometry | within 30 days
  The gross dimensions of resected specimen: length, the distal and proximal resection margins distance, vascular pedicle length
3-year disease free survival | 3 years
  the time from enrollment until disease relapse or death from any cause 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: KeFeng Ding, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No